CLINICAL TRIAL: NCT06261086
Title: Evaluation of Pyroptosis-related Indicators in the Pathogenesis of Vitiligo:Across-sectional Comparative Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Abdelmawla Mohamed, resident of dermatology department at psychatric hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-med-24-01-06MS
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with vitiligo group (Active Comparator): Patients with vitiligo ≥ 18 years old, both male and female patients will be included.
  Exclusion criteria:
  Patients with the following criteria will be excluded from our study:
  1. Pregnancy and breast-feeding women.
  2. patients on antioxidants or anti-inflammatory drugs
  3. Patients on topical/systemic treatment for vitiligo in the last 4weeks prior to enrollment in the study
  4. Patients with other dermatological diseases as psoriasis, lichen planus, viral infection, etc.
  5. Patients suffering from chronic medical illness such as; diabetes mellitus, thyroid disease, and cancer.
  Interventions: Diagnostic Test: evaluate serum levels pyroptosis-related indicators (GASDM-D, IL 1β & IL-18)
- control group (Active Comparator): control criteria with the following criteria will be excluded from our study:
  1- Pregnancy and breast-feeding women.
  Interventions: Diagnostic Test: evaluate serum levels pyroptosis-related indicators (GASDM-D, IL 1β & IL-18)

INTERVENTIONS:
Diagnostic Test: evaluate serum levels pyroptosis-related indicators (GASDM-D, IL 1β & IL-18) — 2 ml blood will be collected from all participants (patients and controls) by aseptic venipuncture into plain tubes. Then the samples will be allowed to coagulate during 10-20 minutes. Serum will be obtained by centrifugation at speed of 2000-3000 cycle/min for 20 minutes. Then we collect the supernatant which immediately be frozen at -80°C until analyzed to determine serum levels of pyroptosis-related indicators (GASDM-D, IL 1β & IL-18). Serum concentration will be assessed by a commercially available double antibody sandwich enzyme-linked immunosorbent assay (ELISA) kit

SUMMARY:
Vitiligo is an acquired pigmentary disorder on skin and/or mucosae, which is characterized by death of melanocytes (MCs), affecting 0.5%-2% of the population worldwide (1). It doesn't affect the health of patients but it has marked social pressure and greatly interfere with their quality of life (2,3). It presents with well circumscribed milky white patches that occur secondary to destruction of melanocyte, it may appear at any age and affect both sexes equally.

It can affect ethnic groups and people of all skin types with no predilection (4).

Clinically, several types of vitiligo are distinguished according to the distribution of the achromic lesions. One or more lesions in a dermatomal pattern are characteristic for segmental vitiligo (SV) while this segmental distribution is absent in non-segmental vitiligo (NSV). The latter variety includes both the focal type and the generalized type (5). Numerous previous studies tried to illustrate the pathogenesis behind the disease, but the exact pathophysiology is still not fully understood. It is a multifactorial disease. Factors include, neural theory, oxidative stress theory, autoimmune hypothesis, intrinsic theory, melanocytorrhagy hypothesis (6). Many theories tried to explain the mechanisms of MC destruction in vitiligo. Apoptosis is one of the most widely studied cell death pathways. In addition, the other two forms of cell death, conventional necrosis and autophagy seem to be involved in the death of vitiligo MCs under certain situations. Moreover, new types of regulated cell death including necroptosis, pyroptosis, and ferroptosis may also participate in the pathogenesis (7). Pyroptosis is a highly inflammatory form of necrosis cell death NCD regulated mainly by caspase-1, which is initiated following large supramolecular complex ermed inflammasome activation (8). The inflammasome-activated Caspases then cleave the pyroptosis-inducing protein Gasdermin D (GSDMD), which forms a pore in the plasma membrane and causes cell lysis as well as the secretion of IL-1β typically (9). Another study suggests that inflammasome activation could be a useful marker for assessing disease progression of vitiligo (10). However, the link between vitiligo and inflammasome activation is still unclear. The inflammasome regulates cell death and inflammation via activation of caspase-1 (11). The activation of caspase-1 promotes the secretion of proinflammatory cytokines IL-1β and IL-18, as well as the initiation of pyroptosis (12). So, evaluation of pyroptosis-related indicators (GASDM-D, IL 1β & IL-18) may help understanding the obscure inflammasome pathway involvement in the pathogenesis of Vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vitiligo ≥ 18 years old, both male and female patients will be included.

Exclusion Criteria:

* Patients with the following criteria will be excluded from our study:

  1. Pregnancy and breast-feeding women
  2. patients on antioxidants or anti-inflammatory drugs
  3. Patients on topical/systemic treatment for vitiligo in the last 4weeks prior to enrollment in the study
  4. Patients with other dermatological diseases as psoriasis, lichen planus, viral infection, etc.
  5. Patients suffering from chronic medical illness such as; diabetes mellitus, thyroid disease, and cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-24 (Estimated); Primary Completion 2024-08-24 (Estimated); Study Completion 2024-08-24 (Estimated)

PRIMARY OUTCOMES:
GASDM-D | 6 months
  Evaluartion of serum level of (GASDM-D) in patients with Vitiligo as well as in control health group. 2- To correlate level of GASDM-D with severity of the disease.
IL 1β | 6 months
  Evaluation of serum level of IL 1β in patients with Vitiligo as well as in control health group 2- To correlate level of IL 1β with severity of the disease.
IL-18 | 6 months
  Evaluation of serum level of IL-18 in patients with Vitiligo as well as in control health group 2- To correlate level of IL-18 with severity of the disease.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kruger C, Schallreuter KU. A review of the worldwide prevalence of vitiligo in children/adolescents and adults. Int J Dermatol. 2012 Oct;51(10):1206-12. doi: 10.1111/j.1365-4632.2011.05377.x. Epub 2012 Mar 27. PMID 22458952
- [Background] Salman A, Kurt E, Topcuoglu V, Demircay Z. Social Anxiety and Quality of Life in Vitiligo and Acne Patients with Facial Involvement: A Cross-Sectional Controlled Study. Am J Clin Dermatol. 2016 Jun;17(3):305-11. doi: 10.1007/s40257-016-0172-x. PMID 26818062
- [Background] Osinubi O, Grainge MJ, Hong L, Ahmed A, Batchelor JM, Grindlay D, Thompson AR, Ratib S. The prevalence of psychological comorbidity in people with vitiligo: a systematic review and meta-analysis. Br J Dermatol. 2018 Apr;178(4):863-878. doi: 10.1111/bjd.16049. Epub 2018 Feb 7. PMID 28991357
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315